CLINICAL TRIAL: NCT04924023
Title: The Effect of Using a Kaleidoscope During Central Venous Catheter Dressing Changes on Anxiety and Pain in Children With Cancer: A Randomised Controlled Study
Brief Title: The Effect of Using a Kaleidoscope During Central Venous Catheter Dressing Changes in Children With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Pınar BEKAR, Assistant Professor, Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KAEK-791
Record Dates: First submitted 2021-06-07; First posted 2021-06-11 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-06

CONDITIONS: Pain; Anxiety
Keywords: Anxiety; Cancer; Central venous catheter; Child; Pain
MeSH Terms: conditions — Pain; Anxiety Disorders; Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomization was done using the closed-envelope method. A total of 60 cards, equally divided between the kaleidoscope and control groups (30 of each), were placed in sealed envelopes. The children were asked to choose one of these envelopes, which determined their placement in the kaleidoscope group or the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kaleidoscope Group (Experimental): Children in this group were told what a kaleidoscope is and how to use it before their central venous catheter dressing. The children were then asked if they would like to look into the kaleidoscope. The children looked into the kaleidoscope and slowly turned it. The researcher asked the children about the colours and shapes seen inside the kaleidoscope. This distraction procedure began immediately before the central venous catheter dressing and continued until it was finished. The kaleidoscope was disinfected before each use. A kaleidoscope was provided for all children in this group by the same researcher. Parents accompanied their children during the catheter dressing.
  Interventions: Behavioral: kaleidoscope application
- Control Group (No Intervention): No intervention was performed to reduce pain and anxiety for children in the control group. Parents accompanied their children during the procedure.

INTERVENTIONS:
Behavioral: kaleidoscope application — The children looked into the kaleidoscope and slowly turned it. The researcher asked the children about the colours and shapes seen inside the kaleidoscope. This distraction procedure began immediately before the central venous catheter dressing and continued until it was finished.
  Arms: Kaleidoscope Group

SUMMARY:
Many medical interventions, including the dressing of central venous catheters, a common procedure used for children with cancer, cause anxiety and pain in children. This can adversely affect their care and recovery. This study aims to determine the effect of using a kaleidoscope during central venous catheter dressing on anxiety and pain in children with cancer.

DETAILED DESCRIPTION:
This was a randomised controlled trial with 60 children aged 6-12 diagnosed with cancer who were placed either in a kaleidoscope group (n=30) or a control group (n=30). Each child's anxiety was evaluated by the child using the Child Fear Scale before, during and after a central venous catheter dressing procedure, and each child's pain during and after the procedure was evaluated by the child using the Wong-Baker Faces Pain Rating Scale (WB-FACES). Each child's heart rate and oxygen saturation were measured with a pulse oximeter device before, during and after central venous catheter dressing.

The children in kaleidoscope group looked into the kaleidoscope and slowly turned it. This distraction procedure began immediately before the central venous catheter dressing and continued until it was finished.

No intervention was performed to reduce pain and anxiety for children in the control group.

Parents accompanied their children during the procedure in both groups.

ELIGIBILITY:
Inclusion Criteria:

* a cancer diagnosis,
* having a central venous catheter,
* 6-12 years old,
* not having taken any analgesics in the 6 hours before the central venous catheter dressing, -being in a non-terminal phase of the disease,
* absence of neutropenia,
* volunteering to participate in the study,
* the absence of any health problems that prevent communication in the parent or the child.

Exclusion Criteria:

-the reporting of pain for another reason at the time of the central venous catheter dressing.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Wong-Baker FACES Pain Rating Scale (WB-FACES) | 5 MONTHS
  The Wong-Baker Faces Pain Rating Scale (WB-FACES) is used to evaluate pain levels in children. This numeric rating scale ranges from 0 to 10 and is represented by faces that display emotions ranging from smiling (0 = very happy or no pain) to crying (10 = the worst pain).
Children's Fear Scale (CFS) | 5 MONTHS
  The Children's Fear Scale (CFS) is used to evaluate anxiety levels in children. It consists of five facial expressions representing a range from no anxiety (0) to severe anxiety (4).

SECONDARY OUTCOMES:
Heart Rate | 5 MONTHS
  The heart rate and oxygen saturation values of the children in both groups were measured and recorded by the researcher 3 minutes before the procedure, during the procedure and 5 minutes after the procedure using a pulse oximeter device.
Oxygen Saturation | 5 MONTHS
  The heart rate and oxygen saturation values of the children in both groups were measured and recorded by the researcher 3 minutes before the procedure, during the procedure and 5 minutes after the procedure using a pulse oximeter device.

CONTACTS AND LOCATIONS:
Overall Officials: Emine EFE, Prof.Dr., Study Director — Akdeniz University, Department of Child Health and Disease Nursing
Locations (1):
- Pınar BEKAR, Burdur, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bekar P, Erkul M, Efe E. The effect of using a kaleidoscope during central venous catheter dressing changes on pain and anxiety in children with cancer: A randomised controlled trial. Eur J Oncol Nurs. 2022 Apr;57:102114. doi: 10.1016/j.ejon.2022.102114. Epub 2022 Feb 25. PMID 35248915